CLINICAL TRIAL: NCT04464278
Title: Predictive Value of Variation in Body Composition on the Fate of Older Subjects During SSR Hospitalization (Suite Care and Rehabilitation)
Brief Title: Variation in Body Composition on the Fate of Older Subjects During SSR Hospitalization
Acronym: VALCOR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR S 1136 (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200265; IDRCB 2019-A03287-50 (Other: ANSM)
Record Dates: First submitted 2020-06-08; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Body Weight Changes
Keywords: Geriatric; Suite Care and Rehabilitation; Body composition
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: weight loss ≥ 5%
- Control group: weight loss ≤ 5%

SUMMARY:
The aim of this study is to correlate weight variation as well as body composition with mortality and unscheduled readmission of geriatric population

DETAILED DESCRIPTION:
Weight loss in obese adults confers health benefits, while weight loss in the elderly is associated with an increased risk of mortality.

There are a large number of studies associating weight loss and mortality but the relationships between changes in body composition (ratio between fat mass and lean mass) and mortality are often contradictory and poorly understood in elderly subject. The aim at this study is to request at this question.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥70 years old
* Hospitalized in SSR for less than 7 days
* No patient opposition

Exclusion Criteria:

* patient with a pacemaker
* lake of nutritional assessment on admission
* lake of assessment of autonomy at admission
* Patient under guardianship or curatorship
* Patient participating in another clinical research
* Patient for whom a short stay (<21 days) is planned in SSR

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric population hospitalized in geriatric department at Rothschild and Emile-Roux hospitals
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The prognosis value of variation of weight on mortality | 3 months
  Determination of variation of weight between D0 and D21 after inclusion
Mortality rate | 3 months
  Monitoring of survival at 3 months after inclusion

SECONDARY OUTCOMES:
The pprognosis value of variation of weight on unscheduled readmission in SSR | Between D0 and D21
  Determination of variation of weight between D0 and D21 after inclusion
Unscheduled readmission in SSR | during 15 days after the end of hospitalization
  Monitoring of unscheduled readmission during 15 days after the end of hospitalization
Lean mass pronostic value | 3 months after the inclusion
  Determine the prognosis value of variation in lean mass on mortality and unscheduled readmission in SSR within 15 days of end of hospitalization
In fat mass pronostic value | 3 months after the inclusion
  Determine the prognosis value of variation in fat mass on mortality and unscheduled readmission in SSR within 15 days of end of hospitalization
fat / lean mass ratio | 3 months after the inclusion
  Determine the prognosis value of fat / lean mass ratio on mortality and unscheduled readmission in SSR within 15 days of end of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Christine FORASASSI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris